CLINICAL TRIAL: NCT05125978
Title: National, Multicenter, Randomized, Double-blind, Triple-dummy, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Canadá Association in the Treatment of Chronic Pain
Brief Title: Efficacy and Safety of Canadá Association in the Treatment of Chronic Pain
Acronym: CANADÁ
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategy review
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1120 - CANADÁ
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Pain, Chronic
Keywords: Analgesia; Pain Management
MeSH Terms: conditions — Chronic Pain; Agnosia | interventions — Dipyrone; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Canadá association (Experimental): The study is triple-dummy, thus the patient must take 3 tablets twice a day, as follows:
  1 tablet Canadá, oral;
  1 placebo tablet of tramadol, oral;
  1 placebo tablet of dipyrone, oral.
  Interventions: Drug: Canadá; Other: Dipyrone placebo; Other: Tramadol hydrochloride placebo
- Tramadol (Active Comparator): The study is triple-dummy, thus the patient must take 3 tablets twice a day, as follows:
  1 tablet tramadol, oral;
  1 placebo tablet of Canadá, oral;
  1 placebo tablet of dipyrone, oral.
  Interventions: Other: Canadá placebo; Other: Dipyrone placebo; Drug: Tramadol hydrochloride
- Dipyrone (Active Comparator): The study is triple-dummy, thus the patient must take 3 tablets twice a day, as follows:
  1 tablet dipyrone, oral;
  1 placebo tablet of tramadol, oral;
  1 placebo tablet of Canadá, oral.
  Interventions: Other: Canadá placebo; Drug: Dipyrone; Other: Tramadol hydrochloride placebo

INTERVENTIONS:
Drug: Canadá — Canadá association 1 tablet twice a day
  Arms: Canadá association
Other: Canadá placebo — Placebo of Canadá association 1 tablet twice a day
  Arms: Dipyrone; Tramadol
Drug: Dipyrone — Dipyrone 1 tablet twice a day
  Arms: Dipyrone
Other: Dipyrone placebo — Placebo of dipyrone 1 tablet twice a day
  Arms: Canadá association; Tramadol
Drug: Tramadol hydrochloride — Tramadol 1 coated tablet twice a day
  Arms: Tramadol
Other: Tramadol hydrochloride placebo — Placebo of tramadol 1 coated tablet twice a day
  Arms: Canadá association; Dipyrone

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Canadá association in the treatment of chronic pain

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the consent form;
* Chronic pain during at least 3 months.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of participants;
* History of alcohol abuse or illicit drug use;
* Participation in a clinical trial in the year prior to this study;
* Pregnancy or risk of pregnacy and lactating participants;
* Known hypersensitivity to any of the formula compounds.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Difference in pain intensity assessed by the VAS scale | 12 weeks
  Change from baseline in the pain intensity escores assessed in medical visits.

SECONDARY OUTCOMES:
Adverse events | 16 weeks
  Incidence and severity of adverse events recorded during the study